CLINICAL TRIAL: NCT00136799
Title: Efficacy and Safety of Fluvastatin in Different Doses in Adults With Mixed Dyslipidemia or Primary Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CXUO320B2302
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Mixed Dyslipidemia; Hypercholesterolemia
Keywords: Mixed Dyslipidemia; high cholesterol; adults; fluvastatin
MeSH Terms: conditions — Hypercholesterolemia | interventions — Fluvastatin

INTERVENTIONS:
Drug: Fluvastatin

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of fluvastatin 80 mg in a Chinese population. This study is not recruiting patients in the US.

ELIGIBILITY:
Inclusion Criteria:

* Mixed dyslipidemia
* Primary hypercholesterolemia

Exclusion Criteria:

* Pregnant or lactating women
* Age > 18 years

Other protocol-defined inclusion and exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2005-06; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in low density lipoprotein cholesterol after 12 weeks

SECONDARY OUTCOMES:
Percent change from baseline in total cholesterol after 12 weeks
Percent change from baseline in high density lipoprotein cholesterol after 12 weeks
Percent change from baseline in total triglycerides after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, Shanghai, China